CLINICAL TRIAL: NCT05776069
Title: A Multi-Modular Trial to Evaluate VGA039 in Healthy Volunteers and Patients With Von Willebrand Disease and Other Bleeding Disorders (VIVID)
Brief Title: Study of VGA039 in Healthy Volunteers and Patients With Von Willebrand Disease (VIVID)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vega Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VGA039-CP001
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Von Willebrand Diseases
Keywords: Von Willebrand Disorder; VWD; Star Therapeutics; Vega Therapeutics; VIVID; VIVID-1; VIVID-2; VIVID-3; VIVID-5; Bleeding disorders; VGA039; Blood coagulation disorders
MeSH Terms: conditions — von Willebrand Diseases; Hemostatic Disorders; Blood Coagulation Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 (Placebo Comparator): Cohorts 1-8 IV or SC VGA039 or Placebo dose to be determined
  Interventions: Drug: VGA039; Other: Placebo
- Part 2 (Experimental): Cohorts A-H IV or SC VGA039 dose to be determined
  Interventions: Drug: VGA039
- Part 3 (Experimental): Cohorts MD-1 to MD-4, SC VGA039 multiple doses, dose to be determined
  Interventions: Drug: VGA039
- Part 4 (Experimental): Cohorts of VGA039 single dose for surgical prophylaxis
  Interventions: Drug: VGA039
- Part 5 (Experimental): Multiple doses of VGA039 in open label extension

INTERVENTIONS:
Drug: VGA039 — Single doses of VGA039
  Arms: Part 1; Part 2; Part 4
Other: Placebo — Single doses of Placebo
  Arms: Part 1
Drug: VGA039 — Multiple doses of VGA039
  Arms: Part 3

SUMMARY:
The VIVID study is structured in a master protocol format comprised of multiple parts that evaluate intravenous (IV) and subcutaneous (SC) VGA039 in healthy volunteers and subjects with von Willebrand Disease (VWD) and other bleeding disorders.

DETAILED DESCRIPTION:
This first-in-human study consists of 5 parts based on the subject population. Part 1 is a randomized, double-blind, placebo-controlled, single-ascending dose (SAD) evaluation of IV or SC VGA039 or placebo in up to 8 cohorts in healthy volunteers. Part 2 is an open-label, SAD of SC or IV VGA039 in up to 8 cohorts in subjects diagnosed with VWD. All participants will be enrolled, treated, and followed up for 15 weeks (IV SAD) or 8 weeks(SC SAD). Part 3 is an open-label, Phase 1b study of SC multiple doses (MD) of VGA039 in up to 4 cohorts. Part 4 is an open-label, Phase 2 study of SC single, surgical prophylaxis (SP) doses of VGA039 administered prior to a minor surgical procedure in subjects diagnosed with VWD in up to 2 cohorts. Part 5 is an open-label extension (OLE) study of SC MD of VGA039 in eligible subjects diagnosed with VWD who have previously participated in a VGA039 interventional trial.

ELIGIBILITY:
Key Inclusion Criteria (All Subjects)

* Subjects, 18 to 60 years of age, inclusive for Parts 1 and 2
* Subjects, 12 to 60 years of age, inclusive for Parts 3 and 5
* No clinically significant laboratory, ECG, or vital signs results.

Additional Key Inclusion Criteria (for Subjects in Part 1 Only) • Body mass index of 18-32 kg/m2

Additional Key Inclusion Criteria (for Subjects in Part 2 Only)

* Subjects with VWD who are symptomatic, defined as having a history of bleeding or bruising.
* Hemoglobin level ≥ 8 g/dL and platelet count ≥ 150 × 109/L at Screening.

Exclusion Key Criteria (All Subjects)

* Use of hormonal contraceptives within 56 days prior to administration of the study drug.
* Subjects with detection of FV Leiden or Prothrombin G20210A mutation, protein C or S deficiency, antithrombin deficiency, or antiphospholipid antibody syndrome at Screening.
* Subjects with other known pro-thrombotic disorders or abnormal findings in any prior laboratory thrombophilia evaluation.
* History of arterial or venous thrombosis, including superficial thrombophlebitis, or embolism.
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular disease, cerebrovascular disease, peripheral vascular disease, or metabolic dysfunction.

Additional Key Exclusion Criterion (Subjects in Part 1 Only)

• Baseline FVIII activity > 150 IU/dL.

Additional Key Exclusion Criteria (Subjects in Parts 2, 3, 4 and 5 Only)

* Baseline FVIII activity > 50 IU/dL.
* Any acute, clinically significant bleeding event requiring surgical or procedural intervention within 7 days prior to receiving study drug.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] | From start of study drug administration until 15 or 8 weeks after IV or SC study drug administration, respectively
  Incidence, nature and severity of adverse events (AEs) and serious adverse events (SAEs), including dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
Plasma Concentrations of single IV and SC doses of VGA039 | From baseline until 15 or 8 weeks after IV or SC study drug administration, respectively
Pharmacodynamics of single IV and SC doses of VGA039 | From baseline until 15 or 8 weeks after IV or SC study drug administration, respectively
Incidence of Anti-drug antibodies to VGA039 | From baseline until 15 or 8 weeks after IV or SC study drug administration, respectively

CONTACTS AND LOCATIONS:
Locations (25):
- United States (10):
  - Orthopedic Institute for Children (UCLA), Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Hemophilia of Georgia Center for Bleeding & Clotting Disorders of Emory, Atlanta, Georgia
  - Science 37, Inc., Morrisville, North Carolina
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Washington Center for Bleeding Disorders, Seattle, Washington
  - Versiti Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin
- Royal Brisbane & Women's Hospital, Queensland Haemophilia Centre, Herston, Queenland, Australia
- Medical University of Vienna, Vienna, Vienna, Austria
- Brazil (3):
  - Centro de Hemoterapia e Hematologia do Rio de Janeiro HEMORIO, Rio de Janeiro, Rio de Janeiro
  - Hemocentro Unicamp, Campinas, São Paulo
  - Hospital das Clinicas - USP Endereco, São Paulo, São Paulo
- Canada (3):
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Queens University, Kingston, Ontario
  - St. Michaels Hospital, Toronto, Ontario
- K J Somaiya Super Speciality Hospital & Research Centre, Sion, Mumbai, India
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, South Africa
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham, Edgbaston
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Royal Free Hospital, London, London
  - Royal London Hospital, Clinical Haematology Research, Whitechapel, London
  - Imperial College Healthcare NHS Trust- Queen Charlotte's & Chelsea Hospital, London

IPD SHARING:
Plan to Share IPD: No